CLINICAL TRIAL: NCT04819347
Title: The Phase 2, Two Arms, One Site, Safety and Antiviral Activity of Combination Therapy With Albuvirtide and 3BNC117 in Virologically Suppressed Subjects With HIV-1 Infection After Analytical Treatment Interruption
Brief Title: Albuvirtide in Combination With 3BNC117 in Virologically Suppressed Subjects With HIV-1 Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Frontier Biotechnologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABT-3BNC117_202
Record Dates: First submitted 2021-03-22; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — albuvirtide; 3BNC117 antibody

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early treatment of infection (Experimental): HIV-1 infected subjects initiated a stable combination antiretroviral therapy (ART) within 6 months of primary HIV infection (PHI), and had plasma HIV-1 RNA <50 copies/mL for at least 12 months.
  Albuvirtide 0.32 g and 3BNC117 2 g every 2 weeks IV infusion for a total of 14 weeks.
  Interventions: Drug: Albuvirtide; Drug: 3BNC117
- Chronic period of infection treatment (Experimental): Chronically HIV-1 infected subjects initiated a stable combination antiretroviral therapy (ART) after 6 months of primary HIV infection (PHI), and had plasma HIV-1 RNA <50 copies/mL for at least 12 months.
  Albuvirtide 0.32 g and 3BNC117 2 g every 2 weeks IV infusion for a total of 14 weeks.
  Interventions: Drug: Albuvirtide; Drug: 3BNC117

INTERVENTIONS:
Drug: Albuvirtide — Long-Acting HIV-1 Fusion Inhibitor (chemically modified peptide targeting HIV-1 gp41)
  Other Names: ABT
Drug: 3BNC117 — Recombinant, fully human mAb of the IgG1κ isotype that specifically binds to HIV-1 gp120.

SUMMARY:
This is a phase 2 study to evaluate the safety and tolerability of combination therapy with Albuvirtide (ABT) and 3BNC117 in virologically suppressed subjects with HIV-1 infection and explore the potential of viral suppression and viral reservoir clearance after analytical treatment interruption (ATI).

DETAILED DESCRIPTION:
This is an open-label, one site study, in which a total of 24 HIV-1 subjects who are virologically suppressed and stable on daily oral combination antiretroviral therapy will be enrolled.

All eligible patients will be switched from daily oral combination antiretroviral regimen to treatment of ABT and 3BNC117 for 14 weeks. There is a two-week overlap of the baseline oral antiretroviral therapy and the ABT-3BNC117 combination regimen at the beginning of the study treatment, and then the oral ART will be interrupted.

The patients will be monitored for viral rebound every two or four weeks following initiation of ABT-3BNC117 combination and will re-initiate an oral antiretroviral regimen if virological rebound is confirmed with plasma HIV-1 RNA levels above 200 copies/ml on two consecutive test.

Pharmacokinetics of ABT and 3BNC117 will be assessed in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age ≥18 years
2. For cohort 1: HIV-1 infected subjects initiated a stable combination antiretroviral therapy (ART) within 6 months of primary HIV infection (PHI), having the document evidence of initial diagnosis of HIV-1 infection and initiation of ART therapy within 6 months of PHI.

   For cohort 2: Chronically HIV-1 infected subjects initiated a stable combination antiretroviral therapy (ART) after 6 months of primary HIV infection (PHI), having the document evidence of initial diagnosis of HIV-1 infection and initiation of ART therapy after 6 months of PHI.
3. Plasma HIV-1 RNA <50 copies/mL for at least 12 months prior to Screening Visit. An exception for a recorded HIV-1 RNA "blip" (e.g., transient HIV-1 RNA >50 copies/mL) can be considered.
4. Plasma HIV-1 RNA <20 copies/mL at Screening Visit.
5. CD4 cell count >500 cells/µL.
6. Laboratory values at Screening of:

   1. Absolute neutrophil count (ANC) ≥0.75×10∧9/L;
   2. Hemoglobin (Hb) ≥105 g/L (male) or ≥95 g/L (female);
   3. Platelets ≥75×10∧9/L;
   4. Serum alanine transaminase (SGPT/ALT) < 2 x upper limit of normal (ULN)
   5. Serum aspartate transaminase (SGOT/AST) < 2 x ULN
   6. Bilirubin (total) <2.5 x ULN unless Gilbert's disease is present or subject is receiving atazanavir in the absence of other evidence of significant liver disease
   7. Creatinine ≤1.5 x ULN
7. Clinically normal resting 12-lead ECG at Screening Visit or, if abnormal, considered not clinically significant by the Principal Investigator.
8. Both male and female patients and their partners of childbearing potential must agree to use accepted methods of contraception.
9. Females of childbearing potential must have a negative serum pregnancy test at Screening visit and negative urine pregnancy test prior to receiving the first dose of study drug.
10. Subjects who have two or more potential alternative antiretroviral treatment regimens.
11. Willing and able to participate in all aspects of the study, including use of IV medication, completion of evaluations, attendance at scheduled clinic visits, and compliance with all protocol requirements as evidenced by providing written informed consent.

Exclusion Criteria:

1. Any active infection or malignancy requiring acute therapy.
2. Hepatitis B infection as manifest by the presence of Hepatitis B surface antigen (HBsAg).
3. Hepatitis C infection as manifest by positive anti-HCV antibody and positive HCV RNA assay at the time of screening.
4. Females who are pregnant, lactating, or breastfeeding, or who plan to become pregnant during the study
5. Unexplained fever or clinically significant illness within 1 week prior to the first study dose
6. Any vaccination within 2 weeks prior to the first study dose.
7. Subjects BMI<20 or >27 kg/m∧2 [BMI＝weight/height∧2].
8. History of Bleeding Disorder or patients on anti-coagulant therapy
9. Participation in an experimental drug trial(s) within 30 days of the Screening Visit
10. Any known allergy or antibodies to the study drug or excipients
11. Treatment with any of the following:

    1. Radiation or cytotoxic chemotherapy with 30 days prior to the screening visit
    2. Receipt of any fusion inhibitor and monoclonal antibody therapy of any kind in the past.
    3. Immunosuppressants within 60 days prior to the Screening Visit
    4. Immunomodulating agents (e.g., interleukins, interferons), hydroxyurea, or foscarnet within 60 days prior to the screening visit
    5. Oral or parenteral corticosteroids within 30 days prior to the Screening Visit. Subjects on chronic steroid therapy > 5 mg/day will be excluded with the following exception:
    6. Subjects on inhaled, nasal, or topical steroids will not be excluded
12. Any other clinical condition that, in the Investigator's judgment, would potentially compromise study compliance or the ability to evaluate safety/efficacy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants (with sustained viral suppression at week 14) with HIV-1 RNA < 50 copies/mL at Week 26 (24 weeks after ATI) | Week 26
  Proportion of participants with HIV-1 RNA < 50 copies/mL at Week 26.

SECONDARY OUTCOMES:
Mean time to virologic rebound (HIV-1 RNA≥200 copies/mL) after ATI | up to 48 weeks
  Mean time to virologic rebound
Proportion of participants without experiencing virologic rebound (HIV-1 RNA<200 copies/mL) at Week 26 (24 weeks after ATI). | Week 26
  Proportion of participants without experiencing virologic rebound
Proportion of participants with HIV-1 RNA < 50 copies/mL at Week 26 (24 weeks after ATI). | Week 26
  Proportion of participants with HIV-1 RNA < 50 copies/mL at Week 26
Mean change in CD4 cell count after ATI | up to 48 weeks
  Mean change in CD4 cell count
Mean change in CD4/CD8 ration after ATI | up to 48weeks
  Mean change in CD4/CD8 ration
Frequency of emergence of new resistance mutations after virologic rebound | up to 48 weeks
  Frequency of emergence of new resistance mutations
Mean time to achieving HIV-1 RNA < 50 copies/mL after experiencing virologic rebound | up to 48 weeks
  Mean time to achieving HIV-1 RNA < 50 copies/mL after experiencing virologic rebound

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Yao, Study Director — Frontier Biotechnologies Inc.
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No